CLINICAL TRIAL: NCT02350517
Title: A Phase II Trial of Recombinant Human Endostatin Injection (Endostar) Combined With Paclitaxel and Nedaplatin as First-line Therapy in Treating Patients With Recurrent or Metastatic Esophageal Cancer
Brief Title: Endostar Combined With Paclitaxel and Nedaplatin in Treating Patients With Recurrent or Metastatic Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhong Li (Other)
Responsible Party: Sponsor-Investigator, Yuhong Li, MD, Ph D, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endo-17
Record Dates: First submitted 2015-01-24; First posted 2015-01-29 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — nedaplatin; endostar protein; Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel+Nedaplatin+Endostar (Experimental): Patients will receive chemotherapy every 3 weeks: Paclitaxel 175mg/m2 IV over 3 hours on Day 4; Nedaplatin 80mg/m2 IV over 1 hours on Day 4; Endostar 3mg/day for 14 days continuous infusion from Day 1 to Day 14.
  Interventions: Drug: Paclitaxel+Nedaplatin+Endostar

INTERVENTIONS:
Drug: Paclitaxel+Nedaplatin+Endostar — Patients will receive chemotherapy every 3 weeks: Paclitaxel 175mg/m2 IV over 3 hours on Day 4; Nedaplatin 80mg/m2 IV over 1 hours on Day 4; Endostar 3mg/day for 14 days continuous infusion from Day 1 to Day 14
  Other Names: Paclitaxl; Nedaplatin; Endostar; Recombinant Human Endostatin Injection

SUMMARY:
This phase Ⅱ study was designed to evaluate the efficacy and safety of endostar combined with paclitaxel and nedaplatin as first-line therapy in treating patients with recurrent or metastatic esophageal squamous cell cancer.

DETAILED DESCRIPTION:
The prognosis of recurrent or metastatic esophageal squamous cell cancer is poor. However, there is still no standard chemotherapy regimen recommended for this disease because of the lack of trails. Currently, anti-angiogenesis therapy had been proved to improve the survival successfully in colorectal cancer, non-small cell lung cancer, breast cancer, glioma and kidney cancer. Recent studies showed that the high level of VEGF was negative correlated with the prognosis of esophageal cancer. Endostar, as a novel endogenous angiogenesis inhibitors, was proved to significantly inhibited the proliferation and metastasis in esophageal cell lines and animal models. A retrospective study also reported the safety and efficacy of the combination therapy of paclitaxel liposome and recombinant human endostatin. Based on the basis above, we designed this phase Ⅱ study to evaluate the efficacy and safety of endostar combined with paclitaxel and nedaplatin as first-line therapy in treating patients with recurrent or metastatic esophageal squamous cell cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients have provided a signed Informed Consent Form
* Age: 18-75 years old
* Histologically confirmed diagnosis of recurrent or metastatic or unresectable advanced esophageal squamous cell carcinoma
* Patients have neither received any palliative chemotherapy nor adjuvant chemotherapy or concurrent chemotherapy with taxane based drugs or large doses cisplatin (cumulative dose ≥ 300mg/m2). The time from the last adjuvant or concurrent chemotherapy to relapse or metastasis should more than 6 months.
* Measurable disease in at least 1 diameter by CT scan or MRI as per RECIST 1.1 criteria; Targeted lesions should not include primary esophageal lesions
* Life expectancy ≥ 3 months
* Karnofsky score ≥70
* Patient has adequate bone marrow and organ function

  * Leukocyte ≥ 3.5 x 10^9/L
  * eAbsolute Neutrophil Count (ANC) ≥ 1.8 x 10^9/L
  * Platelets ≥ 90 x 10^9/L
  * Hemoglobin ≥ 10g/L
* Patient has adequate liver function

  * AST and ALT not more than 2.5 times ULN (not more than 5.0 times ULN if there is liver metastasis)
  * Serum bilirubin ≤ 1.2 x ULN
  * Creatinine ≤ 1.2 times ULN
  * Alkaline phosphatase ≤ 5.0 times ULN
* No serious complications such as active gastrointestinal hemorrhage, perforation, jaundice, gastrointestinal obstruction, non cancerous fever > 38 ℃.
* Patients with effective contraceptive measures
* Expect good compliance

Exclusion Criteria:

* Patients have received radiotherapy in 3 months.
* Patients with relapse recurrent or metastatic lesions in radiated area.
* Patient has received previous treatment with VEGF inhibitors
* Known severe hypersensitivity to the drugs in the experimental chemotherapy or any of the excipients of these products
* Patients without measureable lesions
* Severe systemic disease out of control such as unstable or uncompensated respiratory,cardiac,liver,renal diseases
* Patients with chronic diarrhea
* Patient has a concurrent malignancy or has a malignancy within 5 years of study enrollment (with the exception of nonmelanoma skin cancer or cervical carcinoma in situ
* psychiatric illness including CNS metastases that would prevent the patient from giving informed consent
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | From the date of first drug administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months

SECONDARY OUTCOMES:
Overall survival | From the date of first drug administration until the date of death, assessed up to 36 months
Overall response rate (ORR) | From the date of first drug administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Number of participants with AEs and SAEs as a measure of Safety | Each follow up vist, assessed up to 2 years
  Each follow up visit, assessed up to 3 years. Date will be assessed at each study visiting using NCI CTCAE version 4.0.
Quality of life | Time from day 1 to date of death, assessed up to 3 years
  Quality of life will be assessed at each study visit using EORTC QLQ-C30 and QLQ-OES18

CONTACTS AND LOCATIONS:
Overall Officials: Yu-hong Li, MD, Ph D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China